CLINICAL TRIAL: NCT00918619
Title: Efficacy and Safety of Sangustop® as Haemostatic Agent Versus a Carrier-bound Fibrin Sealant During Liver Resection (ESSCALIVER)
Brief Title: Efficacy and Safety of Sangustop® as Haemostatic Agent Versus a Carrier-Bound Fibrin Sealant During Liver Resection
Acronym: ESSCALIVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-0804
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hemostasis; Liver Surgery
Keywords: randomized,; controlled,; haemostatic agents,; Sangustop,; Tachosil,; liver resection,; haemostasis
MeSH Terms: interventions — TachoSil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sangustop (Experimental)
  Interventions: Device: Sangustop
- Tachosil (Active Comparator)
  Interventions: Drug: Tachosil

INTERVENTIONS:
Device: Sangustop — Application of Sangustop haemostatic agent on resection area
  Other Names: Sangustop®
  Arms: Sangustop
Drug: Tachosil — Application of Tachosil fibrin sealant on resection area
  Other Names: Tachosil®
  Arms: Tachosil

SUMMARY:
This is a multi-centre, patient-blinded, intra-operatively randomised controlled trial. A total of 126 patients planned for an elective liver resection will be enrolled in 9 surgical centres. The primary objective of this study is to show that the collagen based haemostatic device Sangustop® is not inferior to a carrier-bound fibrin sealant (Tachosil®) in achieving haemostasis after hepatic resection.

DETAILED DESCRIPTION:
During liver resection the control of bleeding is a major concern. The liver is predisposed to diffuse bleeding because of its extreme vascularity. Locally applicable agents (haemostats) are in use in order to achieve control over parenchymatic diffuse bleeding from the resection surface and to prevent intraperitoneal complications attributed to bleeding. These haemostats include bone wax, gelatine, collagen, oxidized regenerated cellulose, fibrin sealant glues, and synthetic glues. A composite product with well documented efficacy is Tachosil®. It consists of a collagen fleece carrying the fibrin glue components human fibrinogen and human thrombin. It was shown in a RCT to be superior in obtaining intraoperative haemostasis over argon beamer in liver resection. A new haemostat product is Sangustop®. It is indicated for local haemostasis of capillary bleeding and bleeding of parenchymal organs. Sangustop® is composed of native absorbable collagen fibrils without any blood serum products or any pharmaceutical activity. The felt structure being rich in surface gives a framework for the adhesion of blood platelets, thus provides an additional impetus to clotting. The aim of this study is to show that the new microfibrillar collagen hemostat Sangustop® is not inferior to the carrier-bound fibrin sealant Tachosil® with regards to haemostatic efficacy.

ELIGIBILITY:
Inclusion:

* Age: > 18 years
* Gender: male / female
* Patients with an indication for liver resection (segmental or non-segmental)
* Willing and able to complete the clinical trial procedures, as described in the protocol
* Signed written informed consent to participate in this clinical trial

Exclusion:

* Presence or sequelae of coagulation disorder, liver cirrhosis, Klatskin tumor
* Concurrent participation in another clinical trial with a medical device or medicinal product or with interfering endpoints
* Concurrent or previous therapy with systemic pharmacologic agents promoting blood clotting including but not limited to tranexamix acid, activated factor VII, and aprotinine
* Known allergy or hypersensitivity to a component of the investigational treatments Sangustop® or TachoSil®, to riboflavin or to proteins of bovine origin
* Pregnancy or breast feeding
* Inability to understand the nature and the extent of the trial and the procedures required
* Missing signed written informed consent to participate in the study

Exclusion criteria to be checked during surgery (liver resection):

* Resection area estimated by operating surgeon < 16cm2
* Infected wound area
* Persistant major bleeding after primary haemostasis
* No bleeding after resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with hemostasis 3 minutes after application of the haemostat product | 3 minutes

SECONDARY OUTCOMES:
Time to hemostasis | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wolf O. Bechstein, Prof. Dr., Principal Investigator — University Hospital, Frankfurt am Main, Germany
Locations (8):
- Universitätsklinik für Chirurgie, Medizinische Universität Graz, Graz, Austria
- Germany (7):
  - Charité Campus Virchow, Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Berlin
  - Krankenhaus Nordwest, Klinik für Allgemein-, Viszeral- und Minimal Invasive Chirurgie, Frankfurt
  - Klinikum der J. W. Goethe-Universität, Klinik für Allgemein- und Visceralchirurgie, Frankfurt am Main
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Mainz, Klinik für Allgemein- und Abdominalchirurgie, Mainz
  - Klinikum Großhadern, Ludwig-Maximilians-Universität, München
  - Technische Universität München, Chirurgische Klinik und Poliklinik, München

REFERENCES:
- [Background] Moench C, Bechstein WO, Hermanutz V, Hoexter G, Knaebel HP. Comparison of the collagen haemostat Sangustop(R) versus a carrier-bound fibrin sealant during liver resection; ESSCALIVER-Study. Trials. 2010 Nov 19;11:109. doi: 10.1186/1745-6215-11-109. PMID 21087530
- [Result] Moench C, Mihaljevic AL, Hermanutz V, Thasler WE, Suna K, Diener MK, Seehofer D, Mischinger HJ, Jansen-Winkeln B, Knaebel HP, Bechstein WO. Randomized controlled multicenter trial on the effectiveness of the collagen hemostat Sangustop(R) compared with a carrier-bound fibrin sealant during liver resection (ESSCALIVER study, NCT00918619). Langenbecks Arch Surg. 2014 Aug;399(6):725-33. doi: 10.1007/s00423-014-1203-9. Epub 2014 Jun 1. PMID 24880345
- [Derived] Malik AK, Amer AO, Tingle SJ, Thompson ER, White SA, Manas DM, Wilson C. Fibrin-based haemostatic agents for reducing blood loss in adult liver resection. Cochrane Database Syst Rev. 2023 Aug 8;8(8):CD010872. doi: 10.1002/14651858.CD010872.pub2. PMID 37551841